CLINICAL TRIAL: NCT02230046
Title: A Single-Dose, Open-Label, Randomized, 3-Way Crossover Pivotal Study to Assess the Bioequivalence of 2 Abiraterone Acetate Coated Tablet Formulations With Respect to the Current Commercial Abiraterone Acetate Uncoated Tablet Formulation Under Fasted Conditions in Healthy Male Subjects
Brief Title: Bioequivalence Study of Abiraterone Acetate Coated and Uncoated Tablet Formulations in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR105286; 212082PCR1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Healthy,; Abiraterone Acetate,; Bioequivalence.
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (ABC) (Experimental): Participants will receive a single oral 1000 milligram [mg] dose of abiraterone acetate in all 3 periods under fasted conditions as: Treatment A (current commercial formulation, 4*250 mg uncoated tablets) in Period 1, Treatment B (current commercial formulation, 4*250 mg coated tablets) in Period 2 and Treatment C (new composition, 2*500 mg coated tablets) in Period 3.
  Interventions: Drug: Abiraterone acetate (Treatment A); Drug: Abiraterone acetate (Treatment B)
- Sequence 2 (BCA) (Experimental): Participants will receive a single oral 1000 milligram [mg] dose of abiraterone acetate in all 3 periods under fasted conditions as: Treatment B (current commercial formulation, 4*250 mg coated tablets) in Period 1, Treatment C (new composition, 2*500 mg coated tablets) in Period 2 and Treatment A (current commercial formulation, 4*250 mg uncoated tablets) in Period 3.
  Interventions: Drug: Abiraterone acetate (Treatment A); Drug: Abiraterone acetate (Treatment B)
- Sequence 3 (CAB) (Experimental): Participants will receive a single oral 1000 milligram [mg] dose of abiraterone acetate in all 3 periods under fasted conditions as: Treatment C (new composition, 2*500 mg coated tablets) in Period 1, Treatment A (current commercial formulation, 4*250 mg uncoated tablets) in Period 2 and Treatment B (current commercial formulation, 4*250 mg coated tablets) in Period 3.
  Interventions: Drug: Abiraterone acetate (Treatment A); Drug: Abiraterone acetate (Treatment B)
- Sequence 4 (ACB) (Experimental): Participants will receive a single oral 1000 milligram [mg] dose of abiraterone acetate in all 3 periods under fasted conditions as: Treatment A (current commercial formulation, 4*250 mg uncoated tablets) in Period 1, Treatment C (new composition, 2*500 mg coated tablets) in Period 2 and Treatment B (current commercial formulation, 4*250 mg coated tablets) in Period 3.
  Interventions: Drug: Abiraterone acetate (Treatment A); Drug: Abiraterone acetate (Treatment B)
- Sequence 5 (BAC) (Experimental): Participants will receive a single oral 1000 milligram [mg] dose of abiraterone acetate in all 3 periods under fasted conditions as: Treatment B (current commercial formulation, 4*250 mg coated tablets) in Period 1, Treatment A (current commercial formulation, 4*250 mg uncoated tablets) in Period 2 and Treatment C (new composition, 2*500 mg coated tablets) in Period 3.
  Interventions: Drug: Abiraterone acetate (Treatment A); Drug: Abiraterone acetate (Treatment B)
- Sequence 6 (CBA) (Experimental): Participants will receive a single oral 1000 milligram [mg] dose of abiraterone acetate in all 3 periods under fasted conditions as: Treatment C (new composition, 2*500 mg coated tablets) in Period 1, Treatment B (current commercial formulation, 4*250 mg coated tablets) in Period 2 and Treatment A (current commercial formulation, 4*250 mg uncoated tablets) in Period 3.
  Interventions: Drug: Abiraterone acetate (Treatment A); Drug: Abiraterone acetate (Treatment B)

INTERVENTIONS:
Drug: Abiraterone acetate (Treatment A) — Participants will receive a single oral 1000 mg dose of abiraterone acetate as Treatment A (current commercial formulation, 4*250 mg uncoated tablets) under fasted conditions on Day 1 of period as specified in the protocol.
  Other Names: JNJ-212082
Drug: Abiraterone acetate (Treatment B) — Participants will receive a single oral 1000 mg dose of abiraterone acetate as Treatment B (current commercial formulation, 4*250 mg coated tablets) under fasted conditions on Day 1 of period as specified in the protocol.
  Other Names: JNJ-212082
Drug: Abiraterone acetate (Treatment B) — Participants will receive a single oral 1000 mg dose of abiraterone acetate as Treatment C (new composition, 2*500 mg coated tablets) under fasted conditions on Day 1 of period as specified in the protocol.
  Other Names: JNJ-212082

SUMMARY:
The purpose of this study is to determine the bioequivalence (equivalence of pharmacokinetic parameters) of 2 abiraterone acetate coated tablet formulations with respect to the current commercial abiraterone acetate uncoated tablet formulation under fasted (without eating or drinking) conditions in healthy male participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized (study medication assigned to participants by chance), open-label (all people know the identity of the intervention), single-center, single-dose and 3-way Crossover (the same medications provided to all participants but in different sequence) pivotal study to determine the bioequivalence of 2 abiraterone acetate coated tablet formulations with respect to the current commercial abiraterone acetate uncoated tablet formulation. Approximately 102 healthy male participants will participate in this study. Participants will be randomly assigned to 1 of 6 treatment sequences. The study will consist of 3 parts: Screening Phase (within 21 days before the first study drug administration of the first period), an open-label treatment Phase consisting of 3 single-dose treatment periods (45 days) and follow-up Phase (5 to 7 days after the last study procedure). The total study duration for each participant will be from 45 days to a maximum of 61 days. Participants will receive a single oral 1000 milligram (mg) dose of abiraterone acetate under fasted conditions either as Treatment A (current commercial formulation, uncoated), Treatment B (current commercial formulation, coated) or Treatment C (new composition, coated). Bioequivalence will be primarily evaluated by pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* If sexually active, participants must always use a condom during the study and for 1 week after last intake of study drug. If sexually active with a pregnant woman or woman of child-bearing potential, participants must agree to abstain from intercourse during the study and for 1 week after last intake of study drug. Participants should not donate sperm during the study and for 1 week after receiving the last dose of study drug
* Body mass index (BMI; weight [kilogram(kg)]/height^2 [meter square (m^2)]) between 18.5 and 30.0 kg/m^2, (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participants is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at Screening
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at Screening as specified in the protocol
* Non-smoker, no history of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or participant's verbal report

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participants or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology or clinical chemistry at Screening
* Presence of sexual dysfunction (abnormal libido, erectile dysfunction, etc.) or any medical condition that would affect sexual function
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before the first dose of the study drug is scheduled through study completion
* History of, or a reason to believe a participants has a history of drug or alcohol abuse within the past 5 years

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  The Cmax is the maximum observed plasma concentration of abiraterone acetate.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC [0-last]) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  The AUC (0-last) is the area under the plasma abiraterone acetate concentration-time curve from time zero to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinite Time (AUC [0-infinity]) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  The AUC (0-infinity) is the area under the plasma abiraterone acetate concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma abiraterone acetate concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration (Tmax) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  The Tmax is the time to reach the maximum observed plasma concentration of abiraterone acetate.
Percentage of Area Under the Plasma Concentration-Time Curve Extrapolated From Last Measurable Concentration to Infinite Time (%AUC, ext) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  Percentage of area under the plasma abiraterone acetate concentration-time curve extrapolated from last measurable concentration to infinite time (%AUC, ext) is calculated using formula: ((AUC [0-infinity] minus- AUC [0-last)]/AUC [0-infinity])*100.
Elimination Half-Life (t 1/2, Lambda) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  Elimination half-life (t 1/2, Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda [z]) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  Lambda (z) is the first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time to Last Quantifiable Plasma Concentration (T [last]) of abiraterone acetate | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose on Day 1 of each period
  Time to last quantifiable plasma concentration of abiraterone acetate will be observed.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to follow-up (5 to 7 days after last dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States